CLINICAL TRIAL: NCT01526434
Title: An Open-label, Observational 12-week Study to Assess Health-related Quality of Life and Patient-reported Outcomes in Patients With Rheumatoid Arthritis Treated With Certolizumab Pegol
Brief Title: Health-related Quality of Life and Patient-reported Outcomes in Rheumatoid Arthritis Patients Treated With Certolizumab Pegol
Acronym: SONAR-12
Status: Completed | Type: Observational
Sponsor: UCB Pharma SA (Industry)
Collaborators: ReSearch Pharmaceutical Services, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: RA0053; UCB-CER-2010-01
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Cimzia; Non-interventional; Multicenter; Postmarketing; Local
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Certolizumab Pegol treatment: Patients with RA who begin therapy with Certolizumab Pegol (CZP) will be consecutively included in accordance with the selection criteria. The choice of medical treatment is made independently by the physician before evaluating the possible participation of the patient in the protocol.

SUMMARY:
The main objective is to assess Health-Related Quality of Life (HRQoL) according to physical function, as measured by a specific Questionnaire (Health Assessment Questionnaire), in Rheumatoid Arthritis (RA) patients who begin therapy with subcutaneous Anti-Tumour Necrosis Factor alpha (TNFα) Certolizumab Pegol (CZP).

DETAILED DESCRIPTION:
An open-label, prospective, and post-authorization observational study. This non-interventional study is designed to establish the importance of the measurement of HRQoL data and patient-reported outcomes in clinical practice in patients with RA, and to assess efficacy and safety use of CZP according to the summary of product characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, aged 18 years or older
* Patient has active Rheumatoid Arthritis according to American College of Rheumatology (ACR) criteria with duration ≥ 3 months
* Patient has DAS28 (ESR) > 4.5 and CRP > 1.0 mg/dl at Baseline
* Patient has failed previous Disease Modifying Anti-Rheumatic Drugs (DMARDs) including Methotrexate treatment
* Patient has initiated treatment with subcutaneous anti-Tumour Necrosis Factor alpha (anti-TNFα) CZP, administered every 2 weeks
* Patient has no other prior anti-TNFα treatment (Naïve Patient) or CZP is administered after failure to the first anti-TNFα treatment (First Switch Patient)
* Patient is considered reliable and capable of adhering to the protocol, visit schedule or medication intake according to the judgment of the physician
* Patient has signed and dated a written informed consent form
* The patient's treatment must be within the terms of Summary of Product Characteristics (SmPC)

Exclusion Criteria:

* Patient has a known hypersensitivity to the active substance or to any of the excipients
* Patient has active Tuberculosis or other severe infections such as Sepsis or Opportunistic Infections
* Patient has moderate to severe Heart Failure (New York Heart Association (NHYA) classes III/IV)
* Patient has any medical or psychiatric condition that, in the opinion of the physician, could jeopardize or would compromise the patient's ability to participate in this study or to complete the scheduled questionnaires
* Pregnant women or women of childbearing potential who are not using adequate contraception to prevent pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RA who begin therapy with CZP will be consecutively included in accordance with the selection criteria. The choice of medical treatment is made independently by the physician before evaluating the possible participation of the patient in the study protocol.
  The study will include approximately 105 patients from 20 to 25 sites in Spain.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12 | From Baseline (Week 0) to Week 12
  The HAQ-DI is a measure of function in Rheumatoid Arthritis. There are 20 items in eight categories that represent a comprehensive set of functional activities on a scale from 0 (without difficulty) to 3 (unable to perform without assistance). The category scores are averaged into an overall HAQ-DI from 0 to 3. Scores of 0 to 1 generally represent mild to moderate difficulty, 1 to 2 represent moderate to severe disability, and 2 to 3 indicate severe to very severe disability.
Number of Adverse Drug Reactions (ADRs) during the study (up to 16 weeks) | From Baseline (Week 0) to the end of the Follow-up Period (Week 16)
  An ADR is an Adverse Event for which a causal relationship between the product and the occurrence is suspected.
Number of Serious Adverse Drug Reactions (SADRs) during the study (up to 16 weeks) | From Baseline (Week 0) to the end of the Follow-up Period (Week 16)
  A SADR is a serious Adverse Event for which a causal relationship between the product and the occurrence is suspected.
Number of subjects with at least one Adverse Drug Reaction (ADR) during the study (up to 16 weeks) | From Baseline (Week 0) to the end of the Follow-up Period (Week 16)
  An ADR is an Adverse Event for which a causal relationship between the product and the occurrence is suspected.

SECONDARY OUTCOMES:
Change from Baseline in the Short Form-36 (SF-36) Item Questionnaire Physical Component Summary (PCS) at Week 12 | From Baseline (Week 0) to Week 12
  The SF-36 measures the Health Related Quality of Life (HRQoL). It is a 36-item survey that measures eight domains of health. Four of these domains belong to physical health and four domains to mental health. Domain scores are generated from the SF-36. In addition, two summary scores can also be derived from the SF-36: The Physical Component Summary (PCS) and the Mental Component Summary (MCS).
Change from Baseline in the Short Form-36 (SF-36) Item Questionnaire Mental Component Summary (MCS) at Week 12 | From Baseline (Week 0) to Week 12
  The SF-36 measures the Health Related Quality of Life (HRQoL). It is a 36-item survey that measures eight domains of health. Four of these domains belong to physical health and four domains to mental health. Domain scores are generated from the SF-36. In addition, two summary scores can also be derived from the SF-36: The Physical Component Summary (PCS) and the Mental Component Summary (MCS).
Change from Baseline in Patient's Assessment of Arthritis Pain- Visual Analog Scale (VAS) at Week 12 | From Baseline (Week 0) to Week 12
  VAS ranges from 0 (no pain) to 100 (worst pain).
Change from Baseline in Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) at Week 12 | From Baseline (Week 0) to Week 12
  The DAS28 is used for assessing disease activity in RA. The number of swollen and tender joints will be assessed using 28-joint counts (tender 28 and swollen 28). The ESR is measured in mm/h. In addition the Patient's General Health (GH) is obtained and recorded on a Visual Analog Scale (VAS) of 100 mm. Using this data, the DAS28 [ESR] can be calculated.
Change from Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 12 | From Baseline (Week 0) to Week 12
  ESR is an inflammatory parameter measured in mm/h.
Change from Baseline in the Rheumatoid Factor (RF) at Week 12 | From Baseline (Week 0) to Week 12
  RF is an inflammatory parameter measured in International Units (IU)/ml.
Change from Baseline in Serum C-reactive Protein (CRP) level at Week 12 | From Baseline (Week 0) to Week 12
  CRP is an inflammatory parameter measured in mg/l.
Change from Baseline in the C3 level at Week 12 | From Baseline (Week 0) to Week 12
  C3 is an inflammatory parameter. This measurement includes only subjects for which C3 data are available in the medical history of the subject.
Change from Baseline in the C4 level at Week 12 | From Baseline (Week 0) to Week 12
  C4 is an inflammatory parameter. This measurement includes only subjects for which C4 data are available in the medical history of the subject.
Predictive value of Baseline global ultrasound index in relation to DAS28 at Week 12 | From Baseline (Week 0) to Week 12
Predictive value of Week 6 global ultrasound index in relation to DAS28 at Week 12 | From Week 6 to Week 12
Predictive value of Baseline laboratory data ESR in relation to DAS28 at Week 12 | From Baseline (Week 0) to Week 12
Predictive value of Week 6 laboratory data ESR in relation to DAS28 at Week 12 | From Week 6 to Week 12
Predictive value of Baseline laboratory data CRP in relation to DAS28 at Week 12 | From Baseline (Week 0) to Week 12
Predictive value of Week 6 laboratory data CRP in relation to DAS28 at Week 12 | From Week 6 to Week 12
Predictive value of Baseline laboratory data RF in relation to DAS28 at Week 12 | From Baseline (Week 0) to Week 12
Predictive value of Week 6 laboratory data RF in relation to DAS28 at Week 12 | From Week 6 to Week 12
Predictive value of Baseline Reduced models of ultrasound joint count in relation to DAS28 at Week 12 | From Baseline (Week 0) to Week 12
Predictive value of Week 6 Reduced models of ultrasound joint count in relation to DAS28 at Week 12 | From Week 6 to Week 12
Predictive value of Baseline Reduced models of ultrasound index in relation to DAS28 at Week 12 | From Baseline (Week 0) to Week 12
Predictive value of Week 6 Reduced models of ultrasound index in relation to DAS28 at Week 12 | From Week 6 to Week 12
Change from Baseline in global ultrasound index at Week 6 | From Baseline (Week 0) to Week 6
  Ultrasound assessment by global ultrasound index consists of 24-joint detection and grading (from 0 to 3) of gray-scale synovitis and power doppler synovial signal.
Change from Baseline in global ultrasound index at Week 12 | From Baseline (Week 0) to Week 12
  Ultrasound assessment by global ultrasound index consists of 24-joint detection and grading (from 0 to 3) of gray-scale synovitis and power doppler synovial signal.
Number of injection site reactions during the study (up to 16 weeks) | From Baseline (Week 0) to the end of the Follow-up Period (Week 16)
  Injection site reactions include: erythema, itching, haematoma, pain, swelling or bruising.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (15):
- Spain (15):
  - 11, A Coruña
  - 15, Barcelona
  - 20, Barcelona
  - 4, Barcelona
  - 7, Barcelona
  - 21, Girona
  - 9, Granada
  - 12, León
  - 17, Lleida
  - 18, Lleida
  - 6, Salamanca
  - 10, Seville
  - 14, Tarragona
  - 16, Tarragona
  - 5, Vigo